CLINICAL TRIAL: NCT01876225
Title: Evaluating Pain and Discomfort Associated With Cervical Punch Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Collaborators: THERE ARE NO FUNDING SOURCES TO THE STUDY. (Unknown)
Responsible Party: Principal Investigator, Efraim Siegler, Head of Cervical Clinic, Carmel Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CMC-13-0033-CTIL
Record Dates: First submitted 2013-06-09; First posted 2013-06-12 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-06

CONDITIONS: Pain; Anxiety
Keywords: cervical biopsy; forced cough; pain; VAS scale
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No coughing (No Intervention): Cervical punch biopsy without forced coughing intervention
- coughing (Experimental): Forced coughing during cervical punch biopsy
  Interventions: Behavioral: Forced coughing during cervical punch biopsy

INTERVENTIONS:
Behavioral: Forced coughing during cervical punch biopsy
  Arms: coughing

SUMMARY:
The use of forced coughing during cervical punch biopsy may reduce pain & discomfort associated with the procedure.

DETAILED DESCRIPTION:
Pain and anxiety are associated with many medical procedures performed in ambulatory setting. Colposcopically guided punch biopsies are a standard procedure performed in women with abnormal cervical cytology, as a part of the diagnosis and treatment selection.

Coughing is thought to provide a distraction and to cause a momentarily increase in blood pressure, reducing pain perception.

Therefore, the present study is designed to compare pain associated with cervical punch biopsy and the effect of forced coughing on pain and pain perception.

ELIGIBILITY:
Inclusion Criteria:

- Women undergoing cervical punch biopsy

Exclusion Criteria:

* Women under 18 years old
* Women currently taking prescription pain medications
* Women who consumed pain medication up to 2 hours prior to the scheduled biopsy.
* Women who refuse to take part in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The pain associated with cervical biopsy | 10 minutes
  Evaluating pain during cervical punch biopsy using VAS 0-10 scale.

SECONDARY OUTCOMES:
Length of cervical punch biopsy with and without cough intervention | 10 minutes
  Measurement of procedure length in minutes

OTHER OUTCOMES:
Number of biopsies taken in a single session | 12 minutes
  During the examination, 1 to 3 cervical punch biopsies will be taken, according to colposcopic cervical appearance.

CONTACTS AND LOCATIONS:
Overall Officials: Efraim Siegler, MD, Principal Investigator — Carmel Medical Center
Locations (2):
- Israel (2):
  - Carmel Medical Center, Haifa
  - Lin Medical Center, Haifa